CLINICAL TRIAL: NCT03158857
Title: A Clinical and Pharmacokinetic Study of the Effectiveness of Hepatitis C Treatment (Sofosbuvir+Daclatasvir) in HIV Co-infected and Non HIV Co-infected Patients at the Level of Non-hospital Based Management in Myanmar
Brief Title: Hepatitis C Treatment Study in Myanmar
Status: Withdrawn | Type: Observational
Why Stopped: Long local IRB process to meet with the treatment deadline
Sponsor: Myanmar Oxford Clinical Research Unit (Other)
Collaborators: Myanmar Liver Foundation (Other); Medical Action Myanmar (Other)
Responsible Party: Sponsor
Other Study IDs: OXTREC 3-17
Record Dates: First submitted 2017-05-16; First posted 2017-05-18 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis C
Keywords: Myanmar; HIV
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Dried blood spots for assessment of Hepatitis C genotype
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hepatitis C monoinfection: Sofosbuvir 400 mg tablet once a day + Daclatasvir 60mg tablet once a day
  Patients with evidence of cirrhosis will be offered treatment for 24 weeks, those who are not cirrhotic will be offered 12 weeks of treatment.
  Interventions: Drug: Sofosbuvir 400 mg
- Hepatitis C and HIV co-infection: Sofosbuvir tablet 400 mg once a day + Daclatasvir tablet 90 mg once a day (increased dose in patients receiving efavirenz. Patients on an alternative HIV drug regimen will receive standard dose i.e. 60 mg)
  Patients with evidence of cirrhosis will be offered treatment for 24 weeks, those who are not cirrhotic will be offered 12 weeks of treatment.
  Interventions: Drug: Sofosbuvir 400 mg

INTERVENTIONS:
Drug: Sofosbuvir 400 mg — These drugs are being offered as part of routine care
  Other Names: Daclatasvir 60 mg

SUMMARY:
Hepatitis C is an important health problem in Myanmar affecting around 3% of the population. New drugs have been developed which have transformed the treatment of this disease around the world with very high success rates. Two of these drugs are now registered for use in Myanmar. In this study 200 patients with chronic hepatitis C(100 with HIV co-infection) will be assessed and started on the new treatment. We will observe them and measure treatment effectiveness and tolerability. In 24 patients extra blood samples will be taken for drug measurements to describe the effect of the drugs on patients in Myanmar in more detail.

DETAILED DESCRIPTION:
Data concerning Hepatitis C virus (HCV) prevalence in Myanmar is scarce. Preliminary results of a survey, conducted in 2015 in different areas in Myanmar estimated a seroprevalence of HCV of around 2.65 %, which represents 1.3 million infected patients. Genotype 6 was mostly found in the northern cities and genotype 3 in the southern and western cities of Myanmar. However, treatment options for HCV in Myanmar remain limited currently, including for patients with HIV co-infection who are generally considered high priority given their increased risk for liver disease.

New direct acting antiviral therapies which can achieve high rates of sustained virological response (SVR) (>90%), defined as complete suppression of the virus 12 weeks after completion of antiviral therapy, are becoming increasingly available worldwide.

In Myanmar, in mid-2015, the guideline for the treatment of chronic hepatitis C infection of the Myanmar GI and Liver Society was revised in line with the recent development of Directly Acting Antiviral (DAA) drugs. This observational study will follow the recommendations for patient care presented in this guideline. Two hundred patients with chronic hepatitis C (100 with HIV co-infection) will be recruited in this observational study of routine care with two newly available antiviral drugs (sofosbuvir+ daclatasvir) in two different groups of patients (with and without HIV coinfection) at two centres in Yangon, Myanmar. Their response to treatment will be monitored. In addition a pharmacokinetic study is planned in a subset of patients to characterise any determinants of treatment response or tolerability in patients in Myanmar. This study will be conducted in compliance with the protocol, GCP and the applicable regulatory requirements

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18- years, male or female
2. Willing and able to comply with program assessment, including routine tests, attendance for follow up and compliance with medicine taking.
3. Able to provide written agreement (or witnessed in the case of patients who cannot read and write)
4. Have a diagnosis of hepatitis C (based on a hepatitis C point-of-care test and then confirmed by PCR) with or without HIV

Additional inclusion criteria for PK sub-study

1. HIV well-controlled on current therapy (co-infected patients only)
2. Willing and able to comply with the additional blood sampling in the PK-PD sub-study protocol for the duration of the study

Exclusion Criteria

1. Current pregnancy (pregnancy test to be performed in women of child-bearing age)
2. Previous HCV therapy.
3. HCV PCR negative
4. Patients with significant renal impairment with Cr Cl < 50 ml/min.
5. Known hypersensitivity to any part of the drug regime.
6. Presence of significant comorbidity with life expectancy of less than 12 months.
7. Clinical evidence of decompensated cirrhosis with current or previous episode of ascites, variceal bleed, encephalopathy, and treated hepatocellular cancer (HCC) [Child-Pugh score B or C].
8. Presence of concomitant medical or social situation that would make it difficult for the patient to comply with program protocol or put the patient at additional risk
9. Concomitant medications that cause unacceptable drug-drug interactions. Additional exclusion criteria for PK sub-study

1. Anaemia (Hb <100 mg/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients with hepatitis C attending the clinics of Medical Action Myanmar and the Myanmar Liver Foundation
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
SVR12 | 12 weeks
  Sustained Virological Response 12 weeks after completion of therapy

SECONDARY OUTCOMES:
AEs | 12-24 weeks
  Frequency of adverse events

OTHER OUTCOMES:
Maximum plasma concentration | 2 years
  C max
Area under the curve | 2 years
  AUC
Elimination half-life | 2 years
  t1/2

CONTACTS AND LOCATIONS:
Overall Officials: Ni Ni Tun, MB BS, Principal Investigator — Medical Action Myanmar; MOCRU; Khin Pyone Kyi, MB BS, Principal Investigator — Myanmar Liver Foundation
Locations (1):
- Medical Action Myanmar, Yangon, Burma

IPD SHARING:
Plan to Share IPD: Undecided